CLINICAL TRIAL: NCT07291492
Title: Examining the Relationship Between Health Literacy Level and Functional Outcomes in Patients With Hand and Forearm Injuries
Brief Title: Health Literacy Level and Functional Outcomes in Patients With Hand and Forearm Injuries
Status: Not yet recruiting | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, HANDE USTA, Assistant Professor, Pamukkale University
Other Study IDs: E-60116787-020-789611
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hand Injuries; Forearm Fractures
Keywords: Health Literacy; Functional Outcomes
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hand and/or forearm injuries: Patients aged 18-65 years who voluntarily agreed to participate and who presented with hand and/or forearm injuries
  Interventions: Other: Patients who were referred to the hand rehabilitation unit for hand or forearm injuries will be followed for 12 weeks

INTERVENTIONS:
Other: Patients who were referred to the hand rehabilitation unit for hand or forearm injuries will be followed for 12 weeks — Conventional hand therapy will be applied (edema and scar management, exercises) for 12 weeks.

SUMMARY:
The aim of this study is to examine the association between health literacy, patient-reported outcome measures, and grip strength in a cohort of patients with hand injuries.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* Voluntarily agreed to participate
* Presented with hand and/or forearm injuries

Exclusion Criteria:

* Concomitant shoulder or elbow injuries
* History of surgery due to neurological, rheumatological, or metabolic conditions affecting the entire upper extremity
* Employment in a health-related profession

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were referred to the hand rehabilitation unit for hand or forearm injuries, aged 18-65 years who voluntarily agreed to participate will be included to the study
Sampling Method: Probability Sample
Enrollment: 117 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-03-23 (Estimated); Study Completion 2026-03-23 (Estimated)

PRIMARY OUTCOMES:
European Health Literacy Scale | post-injury 12th week.
  The scale is based on a conceptual framework comprising three health-related domains (treatment, disease prevention, and health promotion) as well as four information-processing stages (accessing, understanding, appraising/decision-making, and applying health information). The instrument contains 47 items rated on a four-point Likert scale.The total score is standardized to range from 0 to 50. Health literacy levels are categorized as follows: (0-25): insufficient, (>25-33): problematic-limited, (>33-42): sufficient, (>42-50): excellent
Michigan Hand Outcomes Questionnaire | post-injury 12th week
  The MHOQ assesses hand and wrist status across six domains: function, activities of daily living, work performance, pain, aesthetics, and patient satisfaction. It consists of 63 items addressing both hands. Each item is scored on a 1-5 scale, and each domain score is converted to a 0-100 scale. Except for the pain domain, higher scores indicate better outcomes
Grip strength | post-injury 12th week
  Grip strength was assessed according to the procedure recommended by the American Society of Hand Therapists. A Jamar dynamometer was used to evaluate gross grip strength. Measurements were performed with the patient seated without elbow support, the arm in adduction and neutral rotation, the elbow flexed at 90°, the forearm in a neutral position, and the wrist positioned in approximately 30° extension. Beginning with the dominant hand, measurements were taken on both sides. The mean value of three trials was recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We may share de-identified IPD upon reasonable request and subject to appropriate data-use agreements, provided that sharing aligns with participant consent and institutional policies.

REFERENCES:
- [Background] Roh YH, Lee BK, Park MH, Noh JH, Gong HS, Baek GH. Effects of health literacy on treatment outcome and satisfaction in patients with mallet finger injury. J Hand Ther. 2016 Oct-Dec;29(4):459-464. doi: 10.1016/j.jht.2016.06.004. Epub 2016 Oct 17. PMID 27765527
- [Background] Roy M, Okrainec K, Novak CB, von Schroeder HP, Urbach DR, McCabe SJ. Universal Measures of Support Are Needed: A Cross-Sectional Study of Health Literacy in Patients with Dupuytren's Disease. Plast Reconstr Surg. 2019 Feb;143(2):350e-358e. doi: 10.1097/PRS.0000000000005209. PMID 30688895
- [Background] Miclau KR, Kwong JW, Tapp E, Mulakaluri A; sALLud Consortium; Shapiro LM. Evaluating the Association Between Health Literacy and Patient-Reported Outcome Measures After Distal Radius Fracture. J Hand Surg Am. 2025 May 9:S0363-5023(25)00163-7. doi: 10.1016/j.jhsa.2025.03.022. Online ahead of print. PMID 40347201
- See also: World Health Organization (WHO). (2016). Health literacy: The solid facts. — https://iris.who.int/handle/10665/326432